CLINICAL TRIAL: NCT01118195
Title: Executive Dysfunction & Suicide: An Exploration Of Risk Factors In Traumatically Brain Injured Veterans
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Beeta Homaifar, VISN 19 MIRECC
Other Study IDs: VA 05-1100
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Traumatic Brain Injury (TBI); Suicidal Behavior
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TBI and Suicidal Behavior
- TBI and No Suicidal Behavior

SUMMARY:
This is a study to learn more about traumatic brain injury (TBI) and suicidal behaviors. The purpose of this research is to find out more about the issues related to these conditions. This study seeks to explore the relationship between executive dysfunction and suicidal behavior in an outpatient population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of traumatic brain injury, history of suicidal behavior.
2. Age 18-74.
3. Currently receiving care through the Eastern Colorado Health Care System (ECHCS) Denver VA TBI Interdisciplinary Team.

Exclusion Criteria:

1. History of other significant neurological disease.
2. Diagnosis of Schizophrenia.
3. Test of Memory Malingering (TOMM) performance lower than 50%.
4. Behavior which could be described as Substance Abuse in the 7 days prior to participation.
5. Current guardianship or mention of recommendation for guardianship in medical chart within the past six months.
6. Inability to read the informed consent document.
7. Inability to adequately respond to questions regarding the informed consent procedure.
8. Significant hearing impairment.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: outpatient veterans with a history of traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)